CLINICAL TRIAL: NCT00843245
Title: Study of Electrical Bioimpedance in Heart Failure Patients Followed at the Heart Failure Unit of the Santa Creu i Sant Pau Hospital.
Brief Title: Study of Electrical Bioimpedance in Heart Failure.
Acronym: BELIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Universitat Politècnica de Catalunya (Other)
Responsible Party: Dr. Antoni Bayés-Genís, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Other Study IDs: ICREC 001-2009
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Heart Failure; Dyspnea
Keywords: Heart Failure; Electric bioimpedance; Body composition; Diagnosis; monitoring; Prognosis; Total body water
MeSH Terms: conditions — Heart Failure; Dyspnea; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum obtained from routine blood test
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- heart failure: Heart failure attending a HF clinic with or without clinical decompensation
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to determine how electrical impedance is modified in relation to extracellular space body fluid retention detected by an electrical bioimpedance method in patients with heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) is a clinical syndrome presenting currently a high prevalence, morbidity and mortality. The lack of sensitivity of symptoms and signs used to make the diagnosis of the exacerbation of HF, and the knowledge in recent years about the relevance to detect congestion before consulting a specialist or go to the emergency department, support the need of more aggressive management of these patients.

Bioimpedance monitoring devices for bioimpedance can provide useful data for the detection of congestion onset and help the decision-making in treatment.

Because patients with heart failure suffer alterations in body composition, mainly due to the amount of extracellular water, the bioimpedance can objectify these variations. In heart failure, bioimpedance has been tested in two studies with small samples of patients estimating total body water. In other studies , the monitoring of intrathoracic impedance has been performed by measurement systems implanted in cardiac defibrillators or in cardiac resynchronization devices. They have proven to be useful for early detection of decompensation in these patients and to detect changes in impedance before the patient begins the clinical manifestations. Furthermore, it has been correlated the detection of decompensation by these devices with significant increases in NT- proBNP (diagnostic and prognostic marker for HF).

The purpose of our study is to observe these changes in impedance from the patient's skin surface and non-invasively.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients > 18 years of age, male or female

Exclusion Criteria:

* Patients treated with renal substitutive treatment such as hemodialysis or peritoneal dialysis
* Patients with automatic implantable devices or pacemakers.
* Patients with metal prosthesis in right side of the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients attended at the Heart Failure Unit of the Hospital de la Santa Creu i Sant Pau
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-04

PRIMARY OUTCOMES:
To identify if electrical bioimpedance analysis is useful for diagnosis, monitoring and prognosis in patients with heart failure. | 18 months

SECONDARY OUTCOMES:
To analyze segmental and whole-body bioimpedance measures in a population of heart failure patients with multi frequency body composition analysis | 18 months
To study the relation between electrical bioimpedance changes with patients' clinical situation (compensated versus decompensated HF) | 18 months
To assess potential correlations between impedance, clinical status, heart failure functional class, and NT-proBNP. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Ribas Pizá, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Piccoli A, Rossi B, Pillon L, Bucciante G. A new method for monitoring body fluid variation by bioimpedance analysis: the RXc graph. Kidney Int. 1994 Aug;46(2):534-9. doi: 10.1038/ki.1994.305. No abstract available. PMID 7967368
- [Background] Albert NM. Bioimpedance to prevent heart failure hospitalization. Curr Heart Fail Rep. 2006 Sep;3(3):136-42. doi: 10.1007/s11897-006-0013-y. PMID 16914106
- [Background] Soderberg M, Hahn RG, Cederholm T. Bioelectric impedance analysis of acute body water changes in congestive heart failure. Scand J Clin Lab Invest. 2001 Apr;61(2):89-94. doi: 10.1080/00365510151097520. PMID 11347985
- [Background] Steele IC, Young IS, Stevenson HP, Maguire S, Livingstone MB, Rollo M, Scrimgeour C, Rennie MJ, Nicholls DP. Body composition and energy expenditure of patients with chronic cardiac failure. Eur J Clin Invest. 1998 Jan;28(1):33-40. doi: 10.1046/j.1365-2362.1998.00245.x. PMID 9502185
- [Background] Yu CM, Wang L, Chau E, Chan RH, Kong SL, Tang MO, Christensen J, Stadler RW, Lau CP. Intrathoracic impedance monitoring in patients with heart failure: correlation with fluid status and feasibility of early warning preceding hospitalization. Circulation. 2005 Aug 9;112(6):841-8. doi: 10.1161/CIRCULATIONAHA.104.492207. Epub 2005 Aug 1. PMID 16061743
- [Background] Luthje L, Vollmann D, Drescher T, Schott P, Zenker D, Hasenfuss G, Unterberg C. Intrathoracic impedance monitoring to detect chronic heart failure deterioration: relationship to changes in NT-proBNP. Eur J Heart Fail. 2007 Jun-Jul;9(6-7):716-22. doi: 10.1016/j.ejheart.2007.03.005. Epub 2007 Apr 25. PMID 17462948
- [Background] Nescolarde L, Rosell-Ferrer J, Gastelurrutia P, Bayes-Genis A, Calpe J, Hernandez R. Comment on "Is bioelectrical impedance vector analysis of value in the elderly with malnutrition and impaired functionality?". Nutrition. 2009 Mar;25(3):370-1; author reply 371-2. doi: 10.1016/j.nut.2008.10.009. Epub 2008 Dec 11. No abstract available. PMID 19084379